CLINICAL TRIAL: NCT02270944
Title: A Phase II, Randomized, Comparative, Observer-Blind, Multi-Center Study Evaluating the Safety and Immunogenicity of the Liquid Formulation of Group B Streptococcus Trivalent Vaccine and of the Lyophilized Formulation of Group B Streptococcus Trivalent Vaccine in Healthy Non-Pregnant Women Aged 18 to 40 Years
Brief Title: Safety and Immunogenicity of the Liquid Formulation of Group B Streptococcus Trivalent Vaccine and of the Lyophilized Formulation of Group B Streptococcus Trivalent Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 205220; V98_21 (Other: Novartis); 2013-003111-22 (EudraCT Number)
Record Dates: First submitted 2014-10-08; First posted 2014-10-22 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Infections, Streptococcal; Streptococcal Infections
Keywords: GBS; vaccine comparability; Group B Strep
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liquid GBS trivalent vaccine (Experimental): Healthy non-pregnant women aged 18-40 years that received a single dose of liquid GBS trivalent vaccine
  Interventions: Biological: GBS Vaccine
- Lyophilized GBS trivalent vaccine (Active Comparator): Healthy non-pregnant women aged 18-40 years that received a single dose of lyophilized GBS trivalent vaccine
  Interventions: Biological: GBS Vaccine

INTERVENTIONS:
Biological: GBS Vaccine — Liquid formulation of a vaccine containing polysaccharide capsules from serotypes Ia, Ib, and III of the Group B Streptococcus
  Arms: Liquid GBS trivalent vaccine
Biological: GBS Vaccine — Lyophilized formulation of a vaccine containing polysaccharide capsules from serotypes Ia, Ib, and III of the Group B Streptococcus
  Arms: Lyophilized GBS trivalent vaccine

SUMMARY:
The purpose of the present study is to assess and compare in healthy non-pregnant women 18 to 40 years of age the safety and immunogenicity of a liquid formulation of Group B Streptococcus (GBS) Trivalent Vaccine (not requiring reconstitution prior to administration), and of the lyophilized formulation of GBS Trivalent Vaccine, administered in non-pregnant and pregnant women in the clinical development program to date.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy females 18-40 years of age, inclusive.
2. Individuals who have given written consent after the nature of the study has been explained according to local regulatory requirements.
3. Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.
4. Individuals who can comply with all study procedures and are available for follow-up.

Exclusion Criteria:

1. Individuals who are pregnant (urine pregnancy test at Study Day 1) or who anticipate becoming pregnant prior to the end of the study, Day 181 Visit.
2. Individuals "of childbearing potential", heterosexually active, and has not used any of the "acceptable contraceptive methods" for at least 2 months prior to study entry and who will not continue to use acceptable contraceptive methods through to the end of the study, Day 181 Visit.

   * Of childbearing potential is defined as status post onset of menarche and not meeting any of the following conditions: menopausal for at least 2 years, status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy, or status after hysterectomy.
   * Acceptable birth control methods are defined as one or more of the following:

   hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring); barrier (condom with spermicide or diaphragm with spermicide) each and every time during intercourse; intrauterine device (IUD); monogamous relationship with vasectomized partner who was vasectomized for at least six months prior to the subject's study entry; or abstinence/no sexual intercourse.
3. Individuals who are nursing (breastfeeding).
4. Individuals who have participated in any clinical trial with another investigational product 30 days prior to first study visit or who intend to participate in another trial prior to the end of the study, Day 181 Visit.
5. Individuals who have had a previous immunization with a vaccine containing Group B Streptococcus antigens.
6. Individuals who receive:

   * live vaccine 30 days prior to study vaccination
   * inactivated vaccines 15 days prior to study vaccination
   * any vaccines within 30 days after study vaccination
   * exception: an inactivated influenza vaccine may be administered up to 7 days prior to study vaccination or 7 days after study vaccination
7. Individuals with a fever (oral temperature ≥ 38°C) within 3 days prior to Study Day 1.
8. Individuals with acute or chronic infection(s) (e.g. requiring systemic antibiotic treatment or antiviral therapy) within 7 days prior to Study Day 1.
9. Individuals with a history of severe allergic reactions after previous vaccination or medication such as anaphylactic shock, asthma, urticaria, or other allergic reaction or hypersensitivity to any vaccine component.
10. Individuals with known or suspected impairment of the immune system including known or suspected HIV infection or HIV-related disease, a history of or an active autoimmune disorder and receipt of immunosuppressive therapy.
11. Long term use of glucocorticoids, including oral or parenteral prednisone ≥ 20 mg/day or equivalent for more than 2 consecutive weeks (or 2 weeks total) within 30 days prior to enrollment. Use of inhaled, intranasal, intra-articular, or topical corticosteroids is allowed.
12. Individuals who have received blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 12 weeks.
13. Individuals with any progressive or severe neurologic disorder, seizure disorder, epilepsy or Guillain-Barré syndrome.
14. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
15. Individuals who are not able to comprehend and to follow all required study procedures for the whole period of the study.
16. Individuals with history or any illness that, in the opinion of the investigator, might interfere with results of the study or pose additional risk to subjects due to participation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1053 (Actual)
Dates: Start 2014-11-20 (Actual); Primary Completion 2015-04-23 (Actual); Study Completion 2015-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (5):
  - GSK Investigational Site, Redding, California
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Salt Lake City, Utah
- Belgium (3):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
- GSK Investigational Site, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below).
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Beran J, Leroux-Roels G, Van Damme P, de Hoon J, Vandermeulen C, Al-Ibrahim M, Johnson C, Peterson J, Baker S, Seidl C, Dreisbach A, Karsten A, Corsaro B, Henry O, Lattanzi M, Bebia Z. Safety and immunogenicity of fully liquid and lyophilized formulations of an investigational trivalent group B streptococcus vaccine in healthy non-pregnant women: Results from a randomized comparative phase II trial. Vaccine. 2020 Apr 3;38(16):3227-3234. doi: 10.1016/j.vaccine.2020.02.085. Epub 2020 Mar 10. PMID 32169390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1053 subjects were enrolled at Belgium, US and Czech Republic sites.
Pre-assignment Details: Among the 1053 subjects enrolled in the study, 3 subjects were randomized but didn't receive the vaccine. The 3 subjects were excluded and didn't start the study.
Period: Overall Study
Arm/Group | Liquid GBS Trivalent Vaccine | Lyophilized GBS Trivalent Vaccine
Started | 529 | 521
Completed | 518 | 516
Not Completed | 11 | 5
Not completed — Lost to Follow-up | 9 | 4
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liquid GBS Trivalent Vaccine | Lyophilized GBS Trivalent Vaccine | Total
Number analyzed (Participants) | 529 | 521 | 1050
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.1 (6.24) | 27.4 (6.05) | 27.2 (6.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 529 | 521 | 1050
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Serotype Ia GBS IgG Levels in Healthy Non-pregnant Women
Description: To evaluate serotype-specific Ia GBS serum IgG antibody levels (anti-Ia) in healthy non-pregnant women when administered with the liquid GBS trivalent vaccine formulation or the lyophilized GBS trivalent vaccine formulation. Antibody concentrations were measured by Enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL).
Time Frame: At Day 31 after a single vaccination
Population: All subjects in the Full Analysis Set immunogenicity population who received the study vaccine, have no major protocol deviation or other reasons to be excluded as defined prior to unblinding & provided evaluable serum samples both before vaccination and at Day 31 in the protocol required windows.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Liquid GBS Trivalent Vaccine | Lyophilized GBS Trivalent Vaccine
Number analyzed (Participants) | 521 | 513
µg/mL | 6.81 [5.54 to 8.37] | 6.66 [5.40 to 8.21]
Statistical Analysis 1: Comparison: Liquid GBS Trivalent Vaccine vs Lyophilized GBS Trivalent Vaccine; To demonstrate the equivalence of the liquid GBS trivalent vaccine formulation to the lyophilized GBS trivalent vaccine formulation for serotypes Ia when administered to healthy non-pregnant women, as measured by geometric mean concentrations (GMC); Test type: Non-Inferiority or Equivalence — To assess the vaccine formulations equivalence, the lower limit of the two-sided 95% confidence interval (CI) for the ratio of GMCs at Day 31 after vaccination must be > 0.5 and the upper limit of the two-sided 95% CI must be < 2.0 (the entire two-sided 95% CI must be contained in the 0.5, 2.0 interval); ANCOVA; Analysis of covariance (ANCOVA) model with vaccine group and center as fixed effects and log10-prevaccination antibody concentration as a covariate; Ratio of GMCs = 1.02, 95% CI 2-sided [0.79 to 1.32]

2. Primary Outcome: Concentration of Serotype III GBS IgG Levels in Healthy Non-pregnant Women
Description: To evaluate serotype-specific III GBS serum IgG antibody levels (anti-III) in healthy non-pregnant women when administered with the liquid GBS trivalent vaccine formulation or the lyophilized GBS trivalent vaccine formulation. Antibody concentrations were measured by Enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL).
Time Frame: At Day 31 after a single vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Liquid GBS Trivalent Vaccine | Lyophilized GBS Trivalent Vaccine
Number analyzed (Participants) | 492 | 489
µg/mL | 2.42 [1.95 to 3.01] | 2.44 [1.95 to 3.04]
Statistical Analysis 1: Comparison: Liquid GBS Trivalent Vaccine vs Lyophilized GBS Trivalent Vaccine; to demonstrate the equivalence of the liquid GBS trivalent vaccine formulation to the lyophilized GBS trivalent vaccine formulation for serotypes III when administered to healthy non-pregnant women, as measured by geometric mean concentrations (GMC); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of GMCs = 0.99, 95% CI 2-sided [0.76 to 1.30]

3. Primary Outcome: Concentration of Serotype Ib GBS IgG Levels in Healthy Non-pregnant Women
Description: To evaluate serotype-specific Ib GBS serum IgG antibody levels (anti-Ib) in healthy non-pregnant women when administered with the liquid GBS trivalent vaccine formulation or the lyophilized GBS trivalent vaccine formulation. Geometric mean concentrations (GMCs) were measured and expressed in micrograms per milliliter (μg/mL). As the singleton ELISA was no longer in use at the time of serotype Ib testing, results were obtained using multiplex immunoassay.
Time Frame: At Day 31 after a single vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Liquid GBS Trivalent Vaccine | Lyophilized GBS Trivalent Vaccine
Number analyzed (Participants) | 483 | 470
µg/mL | 2.94 [2.37 to 3.65] | 3.14 [2.53 to 3.90]
Statistical Analysis 1: Comparison: Liquid GBS Trivalent Vaccine vs Lyophilized GBS Trivalent Vaccine; to demonstrate the equivalence of the liquid GBS trivalent vaccine formulation to the lyophilized GBS trivalent vaccine formulation for serotypes Ib when administered to healthy non-pregnant women, as measured by geometric mean concentrations (GMC); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of GMCs = 0.94, 95% CI 2-sided [0.72 to 1.22]

4. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events (AEs)
Description: Safety was assessed as the number of subjects who reported solicited local and solicited systemic AEs following a single injection with either liquid or lyophilized GBS trivalent vaccine formulations.
Time Frame: From 6 hours through Day 7 post-vaccination
Population: Analyses were evaluated on the Solicited Safety Set (i.e. all subjects in the exposed set with data on post vaccination local or systemic AEs or other signs of reactogenicity). For 3 treated subjects in the Liquid GBS trivalent vaccine group, no safety data were available and for 4 subjects from both groups, no solicited safety data were reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Liquid GBS Trivalent Vaccine | Lyophilized GBS Trivalent Vaccine
Number analyzed (Participants) | 524 | 519
Participants
  Any local AEs | 247 | 229
  Injection site Erythema: number analyzed (Participants) | 522 | 518
  Injection site Erythema | 16 | 9
  Injection site Induration: number analyzed (Participants) | 521 | 519
  Injection site Induration | 17 | 15
  Injection site Ecchymosis: number analyzed (Participants) | 520 | 519
  Injection site Ecchymosis | 1 | 6
  Injection site Pain: number analyzed (Participants) | 520 | 518
  Injection site Pain | 227 | 205
  Injection site Swelling: number analyzed (Participants) | 522 | 519
  Injection site Swelling | 12 | 5
  Injection site Warmth: number analyzed (Participants) | 521 | 517
  Injection site Warmth | 68 | 57
  Chills: number analyzed (Participants) | 519 | 517
  Chills | 64 | 56
  Myalgia: number analyzed (Participants) | 519 | 519
  Myalgia | 75 | 78
  Malaise: number analyzed (Participants) | 519 | 519
  Malaise | 104 | 103
  Nausea: number analyzed (Participants) | 519 | 519
  Nausea | 83 | 77
  Headache: number analyzed (Participants) | 519 | 518
  Headache | 176 | 187
  Fatigue: number analyzed (Participants) | 518 | 518
  Fatigue | 183 | 190
  Rash: number analyzed (Participants) | 519 | 519
  Rash | 18 | 15
  Arthralgia: number analyzed (Participants) | 518 | 518
  Arthralgia | 49 | 53
  Fever (≥38°C): number analyzed (Participants) | 516 | 515
  Fever (≥38°C) | 8 | 7
  Analgesic/antipyrectic use (prevention): number analyzed (Participants) | 521 | 513
  Analgesic/antipyrectic use (prevention) | 2 | 3
  Analgesic/antipyrectic use (treatment): number analyzed (Participants) | 522 | 512
  Analgesic/antipyrectic use (treatment) | 59 | 69
  Any Systemic AEs | 280 | 278

5. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AEs
Description: Safety was assessed as the number of subjects who reported unsolicited AEs following a single injection with either liquid or lyophilized GBS trivalent vaccine formulations.
Time Frame: From Day 1 to Day 181 (end of the study)
Population: Analyses were evaluated on the Unsolicited AEs Safety Set (i.e. all subjects in the exposed set who provided information about post vaccination unsolicited AEs). There were 3 subjects in the Liquid GBS trivalent vaccine group who were treated but for whom no safety data were available.
Measure: Number; unit: Subjects
Arm/Group | Liquid GBS Trivalent Vaccine | Lyophilized GBS Trivalent Vaccine
Number analyzed (Participants) | 526 | 521
Subjects
  Any AEs | 272 | 276
  At least possibly or probably related AEs | 57 | 52
  Medically attended AEs | 165 | 166
  AEs leading to Withdrawal | 0 | 0
  AEs leading to Hospitalization | 5 | 9
  AEs leading to Death | 0 | 0

6. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: Safety was assessed as the number of subjects who reported SAEs following a single injection with either liquid or lyophilized GBS trivalent vaccine formulations.
Time Frame: From Day 1 to Day 181 (end of the study)
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | Liquid GBS Trivalent Vaccine | Lyophilized GBS Trivalent Vaccine
Number analyzed (Participants) | 526 | 521
Subjects
  Serious AEs | 6 | 9
  At least possibly or probably related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and systemic adverse events (AEs) were collected from Day 1 through Day 7 after vaccination. All unsolicited AEs and serious adverse events (SAEs)were collected from Day 1 through Day 181 (end of the study).
Description: The analyses for serious adverse events and other adverse events were performed on the Unsolicited AEs Safety Set. There were 3 subjects in the Liquid GBS trivalent vaccine group who were treated but for whom no safety data were available.
Arm/Group | Liquid GBS Trivalent Vaccine | Lyophilized GBS Trivalent Vaccine
All-Cause Mortality (participants affected / at risk) | 0/526 | 0/521
Serious Adverse Events (participants affected / at risk) | 6/526 | 9/521
Other Adverse Events (participants affected / at risk) | 439/526 | 430/521
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liquid GBS Trivalent Vaccine (N=526) | Lyophilized GBS Trivalent Vaccine (N=521)
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Liquid GBS Trivalent Vaccine (N=526) | Lyophilized GBS Trivalent Vaccine (N=521)
Nausea (Gastrointestinal disorders) | 86 | 81
Chills (General disorders) | 67 | 57
Fatigue (General disorders) | 186 | 194
Injection site erythema (General disorders) | 88 | 84
Injection site haemorrhage (General disorders) | 33 | 38
Injection site induration (General disorders) | 69 | 60
Injection site pain (General disorders) | 238 | 220
Injection site swelling (General disorders) | 42 | 32
Injection site warmth (General disorders) | 73 | 57
Malaise (General disorders) | 105 | 104
Upper respiratory tract infection (Infections and infestations) | 39 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 | 57
Myalgia (Musculoskeletal and connective tissue disorders) | 76 | 80
Headache (Nervous system disorders) | 188 | 208

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.